CLINICAL TRIAL: NCT03899480
Title: Adoptive Transfer of Haploidentical Natural Killer Cells and IL-15 Super Agonist ALT-803 in Human Immunodeficiency Virus (HIV)
Brief Title: Adoptive Transfer of Haploidentical NK Cells and N-803
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDIM-2018-26587
Record Dates: First submitted 2019-03-14; First posted 2019-04-02 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Hiv; HIV Infections; Immune Deficiency
Keywords: Suppressive Antiretroviral Therapy (ART)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Immunologic Deficiency Syndromes | interventions — Cell Count

STUDY DESIGN:
Intervention Model Description: Non-controlled intervention groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Haploidentical Natural Killer Cells (Experimental): Day -7 the subject will undergo inguinal lymph node biopsy & colonoscopy to obtain ileal & rectal biopsies. Blood samples will be obtained. PBMCs will be obtained to sort into CD4 subsets & measure frequencies of HIV RNA & DNA. On Day -1, the donor will undergo apheresis & donor cells will be obtained & incubated overnight. On Day 0 subjects will be infused with N-803 activated NK cells. Subjects will receive 1st dose of N-803 4 hrs after the infusion. Plasma will be obtained at 2, 4 & 12 hrs after. Subjects will return on Days 2, 4, 7, 10, & 14 for blood draw. Subjects will return Days 21 & 42 for blood work & to receive 2 additional doses of N-803, for a total of 3 doses. Subjects will be monitored for toxicity assessment by targeted physical exam & laboratory evaluations on Days 2, 4, 7, 10, 21, & 42. On day 49, we will perform lymph node biopsy & colonoscopy to obtain ileal & rectal tissues. The patient will then be followed until day 100 post infusion.
  Interventions: Biological: Haploidentical Natural Killer (NK) Cells

INTERVENTIONS:
Biological: Haploidentical Natural Killer (NK) Cells — infusion with N-803 activated NK cells

SUMMARY:
This is a pilot therapeutic study of related donor HLA-haploidentical NK-cell based therapy to determine if the treatment is safe and well-tolerated and if there is any measureable impact on virus reservoirs.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV) infection causes profound and often irreversible changes to the adaptive and innate immune system. In the absence of antiretroviral therapy (ART), Cluster of Differentiation (CD)4+ T cells are progressively depleted, CD8+ T cells are often expanded, and much of the immune system is chronically activated. Much of these abnormalities improve during long-term ART, but the system rarely returns to normal. Notably, chronic inflammation persists indefinitely during ART, and is driven by multiple factors, including HIV production (and perhaps replication), irreversible loss of the mucosal integrity and exposure to gut microbes, and an excess burden of other pathogens such as cytomegalovirus (CMV). How the virus and its host interact during effective ART is the focus of intense investigation.

HIV-1 preferentially infects activated memory CD4+ T cells that express the chemokine receptor CCR5, although resting CD4+ T cells, naïve CD4+ T cells and macrophages can also be infected. The majority of infected and activated CD4+ T cells die quickly, but a small fraction reverts to a resting state and persistent indefinitely as the latent reservoir. Because ART blocks all or nearly all new infection events, the reservoir that exists at the time ART is initiated becomes the reservoir that persists for the life of the individual. This memory T cell viral reservoir is maintained during ART by the long half-life of the infected cell, homeostatic proliferation of these cells and perhaps by low levels of persistent viral replication.

The viral reservoir in peripheral blood exists predominantly in those longer-lived memory CD4+ cells endowed with regenerative potential, including memory stem cells, central memory cells and transitional memory. The reservoir also persists in potentially shorter-lived CD4+ T effector cell populations, but whether these cells represent a stable reservoir or one that is constantly being regenerated via proliferation and differentiation is unknown.

"Shock and Kill". One approach to curing HIV infection that has generated broad support in the field is to induce latently infected cells to produce virus (the "shock") while enhancing the ability of the host to clear these virus-producing cells (the "kill"). Histone deacetylase (HDAC) inhibitors have been shown to increase production of HIV-1 RNA and to a lesser degree virus particles from the viral reservoir in vivo. The magnitude of the effect of HDAC inhibitors is modest at best, and as of yet this class of drugs has had no consistent effect on the frequency of cells that harbor replication-competent HIV. Other classes of anti-latency drugs and immunomodulators are therefore being explored for their capacity to stimulate the viral reservoir.

To augment the capacity of the host to eliminate reservoir cells following activation, several immunologic strategies are being explored. These strategies include therapeutic vaccines, monoclonal antibodies, and immune checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Age-18-65
* Stable ART for at least 12 months.
* Screening plasma HIV RNA levels below level of quantification (<40 to <50 copies RNA/mL depending on the assay).
* Screening CD4 count ≥500 cells/µl
* Laboratory tests (Complete Blood Count, Comprehensive Metabolic Panel, Mg, Phosphorus, international normalized ratio/partial thromboplastin time (INR/PTT), Thyroid stimulating hormone (TSH)/T4,) performed within 14 days of infusion of donor NK cells. All laboratory results (unless otherwise specified) must be Grade 1 or normal based on the DAIDS Adverse Event Grading Scale (Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events v2.0)
* Adequate kidney function defined by estimated Glomerular Filtration Rate (CrCl) > 60 ml/min or ml/min/1.73 m2 (≤ grade 2 per DAIDS) and creatinine ≤ 1.5 x ULN
* Pulmonary Function Testing (PFT) must show FEV1 and DLCOcorr > 50% of predicted if subjects have symptomatic or prior known impairment.
* Normal transthoracic echocardiogram
* Ability to be off prednisone and other immunosuppressive drugs for at least 14 days before infusion of cells
* Women of child bearing potential and men with partners of child bearing potential must agree to use effective contraception during therapy and for 4 months after completion of therapy
* Voluntary written consent provided by the subject

Exclusion Criteria:

* Any condition that precludes leukapheresis, lymph node biopsy or colonoscopy with biopsy
* Active infection other than HIV currently requiring systemic antimicrobial therapy
* History of deep vein thrombosis
* Active significant, tissue invasive fungal infection requiring systemic antifungal therapy (dermatologic conditions requiring only topical therapy are allowed).
* Chronic active hepatitis B or C (defined as antibody positive and DNA+ or HepBsAG+).
* Breastfeeding
* Intended modification of antiretroviral therapy in the next 24 weeks
* NYHA (New York Heart Association) Class III or IV heart failure, uncontrollable supraventricular arrhythmias, any history of a ventricular arrhythmia, or other clinical signs of severe cardiac dysfunction
* Symptomatic congestive heart failure, unstable angina pectoris, or Myocardial infarction within 6 months prior to screening
* Marked baseline prolongation of QT/QTc interval (e.g. demonstration of a QTc interval greater than 500 milliseconds)
* On-going chronic systemic corticosteroid use or other immunosuppressive therapy (a history of mild asthma not requiring therapy is eligible and inhaled corticosteroids is allowed. Topical steroids are allowed.)
* Psychiatric illness/social situations that would limit compliance with study requirements
* Previous diagnosis of an autoimmune disease (e.g. rheumatoid arthritis, lupus, inflammatory bowel disease, multiple sclerosis, vasculitis)
* Use of any anticoagulants within the previous 4 weeks.
* Other illness that in the opinion of the investigator would exclude the patient from participating in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | throughout trial participation: 100 days post infusion
  Toxicity and adverse events will be classified according to Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events v2.0. Scale ranges from grade 0 to 4 with a grade of 0 indicating normal signs and symptoms and a grade of 4 indicating potentially life-threatening signs and symptoms. Grade 2, 3, and 4 adverse events will be considered when determining the safety and tolerability of treatment.
CBC; White Blood Cell Count | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. White blood cell count will be evaluated by principle investigator. WBC outside of established clinical reference range (4.5-11.0 k/ul) may indicate adverse treatment reaction. Total occurrence of abnormal CBC results will be used to determine treatment safety and tolerability.
CBC; Red Blood Cell Count | 2, 3, 10, and 21 day post infusion
  Complete blood count will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Red blood cell count will be evaluated by principle investigator. RBC outside established clinical reference range (2.5-5.5 mil/ul) may indicate adverse treatment reaction. Total occurrence of abnormal CBC results will be used to determine treatment safety and tolerability.
CBC; Hemoglobin | 2, 3, 10, and 21 days post infusion
  Complete blood count will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Hemoglobin will be evaluated by principle investigator. Hemoglobin outside established clinical reference range (14-17 g/dl) may indicate adverse treatment reaction. Total occurrence of abnormal hemoglobin results will be used to determine treatment safety and tolerability.
CBC; Hematocrit | 2, 3, 10, and 21 days post infusion
  Complete blood count will be performed at days 2, 3, 10, 21 post infusion. Hematocrit will be evaluated by principle investigator. Hematocrit outside established clinical reference range (42-52%) may indicate adverse treatment reaction. Total occurrence of abnormal hematocrit results will be used to determine treatment safety and tolerability.
CBC; Mean Corpuscular Volume | 2, 3, 10, and 21 days post infusion
  Complete blood count will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. MCV will be evaluated by principle investigator. MCV outside established clinical reference range (84-96 fl.) may indicate adverse treatment reaction. Total occurrence of abnormal MCV results will be used to determine treatment safety and tolerability.
CBC; Mean Corpuscular Hemoglobin | 2, 3, 10, and 21 days post infusion
  Complete blood count will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. MCH will be evaluated by principle investigator. MCH outside established clinical reference range (28-34 pg) may indicate adverse treatment reaction. Total occurrence of abnormal MCH results will be used to determine treatment safety and tolerability.
CBC; Mean Corpuscular Hemoglobin Concentration | 2, 3, 10, and 21 days post infusion
  Complete blood count will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. MCHC will be evaluated by principle investigator. MCHC outside established clinical reference range (33-36 g/dl) may indicate adverse treatment reaction. Total occurrence of abnormal MCHC results will be used to determine treatment safety and tolerability.
CMP; Sodium | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Sodium concentration will be evaluated by principle investigator. Sodium concentration outside established clinical reference range (136-145 mmol/l) may indicate adverse treatment reaction. Total occurrence of abnormal sodium concentration results will be used to determine treatment safety and tolerability.
CMP; Potassium | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Potassium concentration will be evaluated by principle investigator. Potassium concentration outside established clinical reference range (3.5-5.1 mmol/l) may indicate adverse treatment reaction. Total occurrence of abnormal potassium concentration results will be used to determine treatment safety and tolerability.
CMP; Chloride | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Chloride concentration will be evaluated by principle investigator. Chloride concentration outside established clinical reference range (98-107 mmol/l) may indicate adverse treatment reaction. Total occurrence of abnormal chloride concentration results will be used to determine treatment safety and tolerability.
CMP; Glucose | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Glucose concentration will be evaluated by principle investigator. Glucose concentration outside established clinical reference range (70-99 mg/dl) may indicate adverse treatment reaction. Total occurrence of abnormal glucose concentration results will be used to determine treatment safety and tolerability.
CMP; Calcium | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Calcium concentration will be evaluated by principle investigator. Calcium concentration outside established clinical reference range (8.2-10.2 mg/dl) may indicate adverse treatment reaction. Total occurrence of abnormal calcium concentration results will be used to determine treatment safety and tolerability.
CMP; Blood Urea Nitrogen | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. BUN concentration will be evaluated by principle investigator. BUN concentration outside established clinical reference range (6-25 mg/dl) may indicate adverse treatment reaction. Total occurrence of abnormal BUN concentration results will be used to determine treatment safety and tolerability.
CMP; Creatinine | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Creatinine concentration will be evaluated by principle investigator. Creatinine concentration outside established clinical reference range (0.8-1.3 mg/dl) may indicate adverse treatment reaction. Total occurrence of abnormal creatinine concentration results will be used to determine treatment safety and tolerability.
CMP; Alkaline Phosphatase | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Alkaline phosphatase concentration will be evaluated by principle investigator. Alkaline phosphatase concentration outside established clinical reference range (26-137 u/l) may indicate adverse treatment reaction. Total occurrence of abnormal alkaline phosphatase concentration results will be used to determine treatment safety and tolerability.
CMP; Alanine Transaminase | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Alanine transaminase concentration will be evaluated by principle investigator. Alanine transaminase concentration outside established clinical reference range (15-65 u/l) may indicate adverse treatment reaction. Total occurrence of abnormal alanine transaminase concentration results will be used to determine treatment safety and tolerability.
CMP; Aspartate Transaminase | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Aspartate transaminase concentration will be evaluated by principle investigator. Aspartate transaminase concentration outside established clinical reference range (0-37 u/l) may indicate adverse treatment reaction. Total occurrence of abnormal aspartate transaminase concentration results will be used to determine treatment safety and tolerability.
CMP; Total Bilirubin | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Total bilirubin concentration will be evaluated by principle investigator. Total bilirubin concentration outside established clinical reference range (<1.1 mg/dl) may indicate adverse treatment reaction. Total occurrence of abnormal total bilirubin concentration results will be used to determine treatment safety and tolerability.
CMP; Albumin | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Serum albumin will be evaluated by principle investigator. Serum albumin concentration outside established clinical reference range (3.2-4.7 g/dl) may indicate adverse treatment reaction. Total occurrence of abnormal serum albumin concentration results will be used to determine treatment safety and tolerability.
CMP; Total Protein | 2, 3, 10, and 21 days post infusion
  Comprehensive metabolic panel will be performed at days 2, 3, 10, 21 post infusion to aid in the continuous assessment of safety and tolerability throughout the study. Total protein will be evaluated by principle investigator. Total protein concentration outside established clinical reference range (6.4-8.2 g/dl) may indicate adverse treatment reaction. Total occurrence of abnormal total protein concentration results will be used to determine treatment safety and tolerability.

SECONDARY OUTCOMES:
Decrease in HIV reservoirs | 100 days post infusion
  The secondary outcomes in this study are quantities of virus in well-defined anatomical locations (gut and lymph node). These quantities will be determined before and after administration of the NK cells and N-803 therapy based on RNAscope and DNAscope, which are technologies that measure concentration of target RNA and DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Schacker, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller JS, Rhein J, Davis ZB, Cooley S, McKenna D, Anderson J, Escandon K, Wieking G, Reichel J, Thorkelson A, Jorstad S, Safrit JT, Soon-Shiong P, Beilman GJ, Chipman JG, Schacker TW. Safety and Virologic Impact of Haploidentical NK Cells Plus Interleukin 2 or N-803 in HIV Infection. J Infect Dis. 2024 May 15;229(5):1256-1265. doi: 10.1093/infdis/jiad578. PMID 38207119